CLINICAL TRIAL: NCT05007171
Title: Changes in Anthropometric, Biochemical and DNA Damage Parameters After 3-weeks-567-kcal VLCD in Severely Obese Patients With BMI ≥ 35kg/m2
Brief Title: Changes in Anthropometric, Biochemical and DNA Damage Parameters After 3-weeks VLCD in Severely Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Special Hospital for Extended Treatment of Duga Resa (Other Government)
Collaborators: Institute for Medical Research and Occupational Health (Unknown); University of Zagreb (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNAa3WVLCDiBMI-35/22
Record Dates: First submitted 2021-07-16; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Obesity; Weight Loss; DNA Damage
Keywords: Obesity; Very low calorie diet; Alkine comet assay; FPG oxidative comet assay; DNA damage
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Very low calorie diet (Experimental): Use of very low calorie diet in hospital for 3 weeks
  Interventions: Device: Very low calorie diet

INTERVENTIONS:
Device: Very low calorie diet — During 3 weeks in hospital patients will eat prepared very low calorie diet composed of 50-60% complex carbohydrates with low carbo-glycemic index, 20-25% proteins and 25-30% fat

SUMMARY:
Obesity manifest with inflammation, hyperglycaemia and dyslipidaemia. These conditions disturb redox system by generating excessive reactive oxygen species (ROS) and causing oxidative stress (OS) leading to DNA damage. Very low calorie diet (VLCD) have rapid positive effect on weight loss, glucose homeostasis, inflammation and OS. The aim of study is to test the influence of 3-weeks VLCD on anthropometric, biochemical and genomic parameters in class II and III obesity patients.

DETAILED DESCRIPTION:
Obesity is a chronic disease associated with chronic inflammation, insulin resistance, dyslipidemia, oxidative stress and increased risk for type 2 diabetes, cardiovascular disease, stroke and multiple cancer types. Oxidative stress can lead to base lesions of DNA which could be detected with alkine comet assay and its version with use of formamidopyrimidine DNA glycosylase-endonuclease enzyme in fresh or frozen small volume samples. Dietary caloric restriction has beneficial effects on insulin sensitivity, inflammation, oxidative stress and DNA repair. Very low calorie diet (VLCD) data are scarce, especially on the changing levels of DNA damage.This study will assess the effect of a three-week VLCD used in Special Hospital for extended treatment of Duga Resa in individuals with BMI ≥ 35kg/m2 on the level of primary and oxidative DNA damage as well as body composition and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

* body mass index ≥ 35 kg/m2

Exclusion Criteria:

* pregnancy
* actual tumor diseases
* recent diagnostic or treatment exposures to ionizing radiation in the period of one year
* individuals not willing to stay 3 weeks under supervision under full 24 h surveillance from the medical stuff

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
The changes in the body mass index | Baseline, after 3 weeks of VLCD
  Body mass index (kg/m2) is calculated by using measured body weight (kg) with measured body height (m)
The changes in the body fat mass | Baseline, after 3 weeks of VLCD
  Body fat mass (kg) assessed with bioelectrical impedance method
The changes in the skeletal muscle mass | Baseline, after 3 weeks of VLCD
  Skeletal muscle mass (kg) assessed with bioelectrical impedance method
The changes in the percent body fat | Baseline, after 3 weeks of VLCD
  Percent body fat (%) assessed with bioelectrical impedance method
The changes in fasting glucose concentration | Baseline, after 3 weeks of VLCD
  Concentration of glucose (mmol/L)
The changes in urea concentration | Baseline, after 3 weeks of VLCD
  Concentration of urea (mmol/L)
The changes in insulin concentration | Baseline, after 3 weeks of VLCD
  Concentration of insulin (mIU/L)
The changes in HOMA index | Baseline, after 3 weeks of VLCD
  HOMA index is calculated according to the formula: glucose (mmol/L) x insulin (mIU/L)/22.5
The changes in lipid profile | Baseline, after 3 weeks of VLCD
  Concentrations of triglycerides (mmo/L), LDL (mmol/L), HDL (mmol/L) cholesterol (mmol/L)
The changes in inflammation parameters | Baseline, after 3 weeks of VLCD
  Concentration of C-reactive protein (mg/L)
The changes in inflammation parameters | Baseline, after 3 weeks of VLCD
  Concentration of total white blood cell count

SECONDARY OUTCOMES:
The changes in DNA damage assessed with alkaline comet assay | Baseline, after 3 weeks of VLCD
  Values for alkaline comet assay in μm for tale length
The changes in DNA damage assessed with alkaline comet assay | Baseline, after 3 weeks of VLCD
  Values for alkaline comet assay in % for tale intensity
The changes in oxidative DNA damage assessed with FPG comet assay | Baseline, after 3 weeks of VLCD
  Values for FPG comet assay in % for tale intensity

CONTACTS AND LOCATIONS:
Overall Officials: Mirta Milic, PhD, Principal Investigator — Institute for Medical Research and Occupational Health
Locations (1):
- Special Hospital for Extended Treatment of Duga Resa, Duga Resa, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Usman M, Volpi EV. DNA damage in obesity: Initiator, promoter and predictor of cancer. Mutat Res Rev Mutat Res. 2018 Oct-Dec;778:23-37. doi: 10.1016/j.mrrev.2018.08.002. Epub 2018 Aug 17. PMID 30454680
- [Background] Himbert C, Thompson H, Ulrich CM. Effects of Intentional Weight Loss on Markers of Oxidative Stress, DNA Repair and Telomere Length - a Systematic Review. Obes Facts. 2017;10(6):648-665. doi: 10.1159/000479972. Epub 2017 Dec 14. PMID 29237161
- [Background] Wlodarczyk M, Nowicka G. Obesity, DNA Damage, and Development of Obesity-Related Diseases. Int J Mol Sci. 2019 Mar 6;20(5):1146. doi: 10.3390/ijms20051146. PMID 30845725
- [Background] Hart RW, Dixit R, Seng J, Turturro A, Leakey JE, Feuers R, Duffy P, Buffington C, Cowan G, Lewis S, Pipkin J, Li SY. Adaptive role of caloric intake on the degenerative disease processes. Toxicol Sci. 1999 Dec;52(2 Suppl):3-12. doi: 10.1093/toxsci/52.2.3. PMID 10630584
- [Background] Heydari AR, Unnikrishnan A, Lucente LV, Richardson A. Caloric restriction and genomic stability. Nucleic Acids Res. 2007;35(22):7485-96. doi: 10.1093/nar/gkm860. Epub 2007 Oct 16. PMID 17942423
- [Background] Setayesh T, Nersesyan A, Misik M, Ferk F, Langie S, Andrade VM, Haslberger A, Knasmuller S. Impact of obesity and overweight on DNA stability: Few facts and many hypotheses. Mutat Res Rev Mutat Res. 2018 Jul-Sep;777:64-91. doi: 10.1016/j.mrrev.2018.07.001. Epub 2018 Jul 11. PMID 30115431
- [Background] Setayesh T, Misik M, Langie SAS, Godschalk R, Waldherr M, Bauer T, Leitner S, Bichler C, Prager G, Krupitza G, Haslberger A, Knasmuller S. Impact of Weight Loss Strategies on Obesity-Induced DNA Damage. Mol Nutr Food Res. 2019 Sep;63(17):e1900045. doi: 10.1002/mnfr.201900045. Epub 2019 Jun 14. PMID 31141317
- [Background] Harper C, Maher J, Grunseit A, Seimon RV, Sainsbury A. Experiences of using very low energy diets for weight loss by people with overweight or obesity: a review of qualitative research. Obes Rev. 2018 Oct;19(10):1412-1423. doi: 10.1111/obr.12715. Epub 2018 Aug 24. PMID 30144269
- [Background] Parretti HM, Jebb SA, Johns DJ, Lewis AL, Christian-Brown AM, Aveyard P. Clinical effectiveness of very-low-energy diets in the management of weight loss: a systematic review and meta-analysis of randomized controlled trials. Obes Rev. 2016 Mar;17(3):225-34. doi: 10.1111/obr.12366. Epub 2016 Jan 18. PMID 26775902
- [Background] Milic M, Ozvald I, Vinkovic Vrcek I, Vucic Lovrencic M, Orescanin V, Bonassi S, Del Castillo ER. Alkaline comet assay results on fresh and one-year frozen whole blood in small volume without cryo-protection in a group of people with different health status. Mutat Res Genet Toxicol Environ Mutagen. 2019 Jul;843:3-10. doi: 10.1016/j.mrgentox.2019.03.009. Epub 2019 Mar 28. PMID 31421735
- [Background] Milic M, Kisan M, Rogulj D, Radman M, Lovrencic MV, Konjevoda P, Domijan AM. Level of primary DNA damage in the early stage of metabolic syndrome. Mutat Res Genet Toxicol Environ Mutagen. 2013 Dec 12;758(1-2):1-5. doi: 10.1016/j.mrgentox.2013.07.013. Epub 2013 Sep 27. PMID 24076402
- [Background] Rogulj D, Konjevoda P, Milic M, Mladinic M, Domijan AM. Fatty liver index as an indicator of metabolic syndrome. Clin Biochem. 2012 Jan;45(1-2):68-71. doi: 10.1016/j.clinbiochem.2011.10.014. Epub 2011 Oct 26. PMID 22056738
- [Background] Langie SA, Azqueta A, Collins AR. The comet assay: past, present, and future. Front Genet. 2015 Aug 13;6:266. doi: 10.3389/fgene.2015.00266. eCollection 2015. No abstract available. PMID 26322077
- [Background] Mulligan AA, Luben RN, Bhaniani A, Parry-Smith DJ, O'Connor L, Khawaja AP, Forouhi NG, Khaw KT; EPIC-Norfolk FFQ Study. A new tool for converting food frequency questionnaire data into nutrient and food group values: FETA research methods and availability. BMJ Open. 2014 Mar 27;4(3):e004503. doi: 10.1136/bmjopen-2013-004503. PMID 24674997
- [Background] Heilbronn LK, de Jonge L, Frisard MI, DeLany JP, Larson-Meyer DE, Rood J, Nguyen T, Martin CK, Volaufova J, Most MM, Greenway FL, Smith SR, Deutsch WA, Williamson DA, Ravussin E; Pennington CALERIE Team. Effect of 6-month calorie restriction on biomarkers of longevity, metabolic adaptation, and oxidative stress in overweight individuals: a randomized controlled trial. JAMA. 2006 Apr 5;295(13):1539-48. doi: 10.1001/jama.295.13.1539. PMID 16595757
- [Background] Snel M, Jonker JT, Hammer S, Kerpershoek G, Lamb HJ, Meinders AE, Pijl H, de Roos A, Romijn JA, Smit JW, Jazet IM. Long-term beneficial effect of a 16-week very low calorie diet on pericardial fat in obese type 2 diabetes mellitus patients. Obesity (Silver Spring). 2012 Aug;20(8):1572-6. doi: 10.1038/oby.2011.390. Epub 2012 Jan 26. PMID 22282049
- [Background] Portnay GI, O'Brian JT, Bush J, Vagenakis AG, Azizi F, Arky RA, Ingbar SH, Braverman LE. The effect of starvation on the concentration and binding of thyroxine and triiodothyronine in serum and on the response to TRH. J Clin Endocrinol Metab. 1974 Jul;39(1):191-4. doi: 10.1210/jcem-39-1-191. No abstract available. PMID 4835133
- [Derived] Ozvald I, Bozicevic D, Duh L, Vinkovic Vrcek I, Domijan AM, Milic M. Changes in anthropometric, biochemical, oxidative, and DNA damage parameters after 3-weeks-567-kcal-hospital-controlled-VLCD in severely obese patients with BMI >/= 35 kg m-2. Clin Nutr ESPEN. 2022 Jun;49:319-327. doi: 10.1016/j.clnesp.2022.03.028. Epub 2022 Mar 26. PMID 35623833